CLINICAL TRIAL: NCT06326216
Title: Determination of Baseline Levels for Prostate Cancer-Derived Extracellular Vesicles Following Local Treatment of Prostate Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 19-011292; NCI-2023-05221 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-011292 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — With permission of participant, blood and urine samples may be retained for use in future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Observational (Cohort I): Prostate cancer patients undergo blood and urine sample collection on study. Patients' medical records are also reviewed.
  Interventions: Other: Non-Interventional Study
- Observational (Cohort III): Female urology clinic patients and female volunteers undergo blood and urine sample collection on study.
  Interventions: Other: Non-Interventional Study
- Observational (Cohort II): Prostate cancer patients undergo blood and urine sample collection throughout the study. Patients' medical records are also reviewed.

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Groups: Observational (Cohort I); Observational (Cohort III)

SUMMARY:
This study is being done to determine whether levels of prostate cancer derived extracellular vesicles from blood and urine specimens correlate with response to primary local treatment (surgery) in prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the levels of prostate cancer-derived extracellular vesicles pre- and post-RP.

II. Determine the correlation between levels of prostate cancer-derived extracellular vesicles and PSA.

OUTLINE: This is an observational study. Participants are assigned to 1 of 2 cohorts.

COHORT I (RADICAL PROSTATECTOMY): Prostate cancer patients undergo blood and urine sample collection on study. Patients' medical records are also reviewed.

COHORT II (NEOADJUVANT): Prostate cancer patients undergo blood and urine sample collection throughout the study. Patients' medical records are also reviewed.

COHORT III (NEGATIVE CONTROLS): Female urology clinic patients and female volunteers undergo blood and urine sample collection on study.

ELIGIBILITY:
Inclusion Criteria:

* PROSTATE CANCER PATIENTS:

  * Age 18+
  * Able to give informed consent
  * Patients with prostate cancer
  * Patients treated with primary prostatectomy

    * The focus will be on high-risk patients with at least one of either criterion:
  * PSA >= 20 ng/ml
  * AND/OR Gleason >= 8
  * AND/OR clinical stage >= T3
* FEMALE CONTROL PATIENTS:

  * Age 18+
  * Able to give informed consent

Exclusion Criteria:

* PROSTATE CANCER PATIENTS:

  * Unable or unwilling to provide informed consent
  * Metastatic prostate cancer - defined evidence of metastatic disease on pre-procedural testing
* FEMALE CONTROL PATIENTS:

  * Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer and undergoing prostatectomy as a local treatment and female patients seen in the Urology Clinic or female research volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Levels of prostate cancer-derived extracellular vesicles (EVs) - radical prostatectomy | Pre-surgery; once post-surgery, 6 weeks to 6 months after surgery (likely collected during routine visits); annual blood collection (optional)
  Levels of prostate cancer-derived EVs will be assessed using blood and urine samples
Levels of prostate cancer-derived extracellular vesicles (EVs) - negative controls | Baseline
  Levels of prostate cancer-derived EVs will be assess using blood and urine samples
Correlation between prostate specific antigen (PSA) levels and prostate cancer-derived EVs | Baseline
  PSA levels and EVs will be determined from blood and urine samples and will be assessed by correlation analysis.
Prostate cancer-derived EV levels | Baseline
  Prostate cancer-derived EV levels will be determined from blood and urine samples and will be assessed by comparative analysis between prostate cancer patients and female patients (negative controls).

CONTACTS AND LOCATIONS:
Overall Officials: Eugene D. Kwon, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials